CLINICAL TRIAL: NCT01508117
Title: A Phase II Window Study of Front-line Axitinib Followed by Axitinib and Radiation for Elderly Patients With Glioblastoma Multiforme (GBM)
Brief Title: Phase II Axitinib (AG-013736) in Elderly Glioblastoma Multiforme (GBM) Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: transferred study sponsor
Sponsor: University of Cincinnati (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Rekha Chaudhary, Adjunct Assistant Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCR-2
Record Dates: First submitted 2012-01-06; First posted 2012-01-11 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2014-12

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; brain tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Axitinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib + Radiation Therapy (Experimental): Axitinib 5mg twice daily for 28 days followed by concurrent axitinib plus hypofractionated radiation therapy (45 Gy in 15 fractions) followed by maintenance axitinib 5mg twice daily until progression or unacceptable toxicity
  Interventions: Drug: Axitinib; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Axitinib — 5 mg twice daily starting 21 days after resection and continuing until progression or unacceptable toxicity
  Other Names: AG-013736
Radiation: Radiation Therapy — 45 Gy in 15 fractions starting after 28 days of Axitinib monotherapy
  Other Names: Hypofractionated radiation therapy

SUMMARY:
The purpose of this study is to determine whether the addition of an investigational medication, axitinib, to radiation therapy will improve the outcome of treatment in patients, above the age of 70.

DETAILED DESCRIPTION:
The addition of axitinib to standard treatment is experimental and has not been approved by the United States Food and Drug Administration (FDA). Axitinib works by preventing new blood vessels from forming, and tumors need to make new blood vessels in order to grow. The study will find out what effects, good or bad, axitinib has on the tumor. In addition, this study will try to determine whether the response to axitinib and the overall outcome depends on certain characteristics of your tumor.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with histologically proven glioblastoma multiforme
* Age above 70 years
* Karnofsky score of 50-80
* Adequate organ function as defined by laboratory values
* Life expectancy of >12 weeks
* No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure readings must be 140 mm Hg, and the baseline diastolic blood pressure readings must be 90 mm Hg. Patients whose hypertension is controlled by antihypertensive therapies are eligible.

Exclusion Criteria:

* Prior treatment with chemotherapy or radiation for glioblastoma multiforme
* Patients with extensive tumor hemorrhage
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack and 6 months for deep vein thrombosis or pulmonary embolism

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rekha Chaudhury, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 8/10/11-10/26/12
Period: Overall Study
Arm/Group | Axitinib + Radiation Therapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib + Radiation Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: average 1 year
Measure: Number; unit: years
Arm/Group | Axitinib + Radiation Therapy
Number analyzed (Participants) | 1
years | 0.2

ADVERSE EVENTS:
Time Frame: Duration of treatment
Arm/Group | Axitinib + Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib + Radiation Therapy (N=1)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib + Radiation Therapy (N=1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to lack of accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes